CLINICAL TRIAL: NCT05407675
Title: A Phase 1/2 Study of BMS-986408 Alone and in Combination With Nivolumab or With Nivolumab and Ipilimumab in Participants With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Tolerability of BMS-986408 Alone and in Combination With Nivolumab or Nivolumab and Ipilimumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA099-003
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Oncology; Phase 1; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; Ipilimumab; Paclitaxel; Pemetrexed; Cisplatin; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: BMS-986408 Monotherapy (Experimental)
  Interventions: Drug: BMS-986408
- Part 2: BMS-986408 in combination with nivolumab (Experimental)
  Interventions: Drug: BMS-986408; Biological: Nivolumab
- Part 2: BMS-986408 in combination with nivolumab and ipilimumab (Experimental)
  Interventions: Drug: BMS-986408; Biological: Nivolumab; Biological: Ipilimumab
- Part 2: BMS-986408 in combination with nivolumab and chemotherapy (Experimental)
  Interventions: Drug: BMS-986408; Biological: Nivolumab; Biological: Platinum-doublet chemotherapy
- Part 2: BMS-986408 in combination with rabeprazole (Experimental)
  Interventions: Drug: BMS-986408; Drug: Rabeprazole
- Part 3: BMS-986408 in combination with nivolumab (Experimental)
  Interventions: Drug: BMS-986408; Biological: Nivolumab
- Part 3: BMS-986408 in combination with nivolumab and chemotherapy (Experimental)
  Interventions: Drug: BMS-986408; Biological: Nivolumab; Biological: Platinum-doublet chemotherapy

INTERVENTIONS:
Drug: BMS-986408 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part 2: BMS-986408 in combination with nivolumab; Part 2: BMS-986408 in combination with nivolumab and chemotherapy; Part 2: BMS-986408 in combination with nivolumab and ipilimumab; Part 3: BMS-986408 in combination with nivolumab; Part 3: BMS-986408 in combination with nivolumab and chemotherapy
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Part 2: BMS-986408 in combination with nivolumab and ipilimumab
Biological: Platinum-doublet chemotherapy — Specified dose on specified days
  Other Names: PDCT; carbplatin, paclitaxel, pemetrexed, cisplatin
  Arms: Part 2: BMS-986408 in combination with nivolumab and chemotherapy; Part 3: BMS-986408 in combination with nivolumab and chemotherapy
Drug: Rabeprazole — Specified dose on specified days
  Arms: Part 2: BMS-986408 in combination with rabeprazole

SUMMARY:
The primary purpose of this study is to characterize the safety profile of BMS-986408 as monotherapy and in combination with nivolumab or nivolumab and ipilimumab to establish the maximum tolerated dose (MTD). The Recommended Phase 2 Dose (RP2D) that optimizes the pharmacokinetic/pharmacodynamic (PK/PD) relationship of BMS-986408 will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a histologically or cytologically confirmed, advanced, unresectable/metastatic, solid malignancy of any histology measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Participants who have received, been refractory to, ineligible for, or intolerant of existing therapy(ies) known to provide clinical benefit for the condition of the participant
* Participants with melanoma should have documentation of mutation status for B-type Raf proto-oncogene (BRAF) and neuroblastoma ras viral oncogene homolog (NRAS)
* Participants must have experienced radiographically documented progressive disease on or after the most recent therapy

Exclusion Criteria:

* An active, known or suspected autoimmune disease
* Conditions requiring systemic treatment with either corticosteroids within 14 days or other immunosuppressive medications within 30 days of the first dose of study treatment
* Current or recent gastrointestinal disease or gastrointestinal surgery that could impact the absorption of study drug
* Untreated central nervous system (CNS) metastases or leptomeningeal metastasis

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (3):
  - Local Institution - 0010, Boston, Massachusetts
  - Local Institution - 0001, Hackensack, New Jersey
  - Local Institution - 0003, Houston, Texas
- Canada (4):
  - Local Institution - 0007, Edmonton, Alberta
  - Local Institution - 0011, Hamilton, Ontario
  - Local Institution - 0005, Ottawa, Ontario
  - Local Institution - 0006, Toronto, Ontario
- France (4):
  - Local Institution - 0015, Bordeaux, Aquitaine
  - Local Institution - 0014, Villejuif, Paris
  - Local Institution - 0018, Marseille
  - Local Institution - 0019, Toulouse
- Spain (4):
  - Local Institution - 0024, Málaga, Andalusia
  - Local Institution - 0025, Madrid, Madrid, Comunidad de
  - Local Institution - 0022, Madrid
  - Local Institution - 0023, Madrid
- Switzerland (3):
  - Local Institution - 0021, Sankt Gallen, Canton of St. Gallen
  - Local Institution - 0012, Basel
  - Local Institution - 0020, Geneva

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not enrolled in Part 3.
Groups:
- Part 1 (Group A) BMS-986408 0.75 mg QD: Participants with advanced solid tumors received 0.75 mg tablets of BMS-986408 once daily (QD).
- Part 1 (Group A) BMS-986408 1.5 mg QD: Participants with advanced solid tumors received 1.5 mg tablets of BMS-986408 once daily (QD).
- Part 1 (Group A) BMS-986408 3 mg QD: Participants with advanced solid tumors received 3 mg tablets of BMS-986408 once daily (QD).
- Part 1 (Group A) BMS-986408 5 mg QD: Participants with advanced solid tumors received 5 mg tablets of BMS-986408 once daily (QD).
- Part 1 (Group A) BMS-986408 7.25 mg QD: Participants with advanced solid tumors received 7.25 mg tablets of BMS-986408 once daily (QD).
- Part 1 (Group B) BMS-986408 1.5 mg BID: Participants with advanced solid tumors received 1.5 mg tablets of BMS-986408 twice in a day (BID).
- Part 1 (Group B) BMS-986408 2.25 mg BID: Participants with advanced solid tumors received 2.25 mg tablets of BMS-986408 twice in a day (BID).
- Part 1 (Group B) BMS-986408 3.75 mg BID: Participants with advanced solid tumors received 3.75 mg tablets of BMS-986408 twice in a day (BID).
- Part 1 Group C BMS-986408 3 mg QD: Participants with advanced, unresectable/metastatic solid malignancy of the following histologies: HNSCC, NSCLC, melanoma, or RCC, have previously received therapy containing anti-PD-1, anti-PD-L1 or anti-CTLA-4 agents, and had received, were refractory to, ineligible for, or intolerant of existing therapies known to provide clinical benefit received 3 mg tablets of BMS-986408 once daily (QD).
- Part 1 Group C BMS-986408 5 mg QD: Participants with advanced, unresectable/metastatic solid malignancy of the following histologies: HNSCC, NSCLC, melanoma, or RCC, have previously received therapy containing anti-PD-1, anti-PD-L1 or anti-CTLA-4 agents, and had received, were refractory to, ineligible for, or intolerant of existing therapies known to provide clinical benefit received 5 mg tablets of BMS-986408 once daily (QD).
- Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W: Participants with advanced, unresectable/metastatic solid malignancy of the following histologies: HNSCC, NSCLC, melanoma, or RCC, have previously received therapy containing anti-PD-1, anti-PD-L1 or anti-CTLA-4 agents, and had received, were refractory to, ineligible for, or intolerant of existing therapies known to provide clinical benefit received 1.5 mg tablets of BMS-986408 once daily (QD) and 480 mg intravenous infusion (approx. 30 minutes) once in 4 weeks (Q4W).
- Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W: Participants with advanced, unresectable/metastatic solid malignancy of the following histologies: HNSCC, NSCLC, melanoma, or RCC, have previously received therapy containing anti-PD-1, anti-PD-L1 or anti-CTLA-4 agents, and had received, were refractory to, ineligible for, or intolerant of existing therapies known to provide clinical benefit received 3 mg tablets of BMS-986408 once daily (QD) and 480 mg intravenous infusion (approx. 30 minutes) once in 4 weeks (Q4W).
- Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W: Participants with advanced, unresectable/metastatic solid malignancy of the following histologies: HNSCC, NSCLC, melanoma, or RCC, have previously received therapy containing anti-PD-1, anti-PD-L1 or anti-CTLA-4 agents, and had received, were refractory to, ineligible for, or intolerant of existing therapies known to provide clinical benefit received 5 mg tablets of BMS-986408 once daily (QD) and 480 mg intravenous infusion (approx. 30 minutes) once in 4 weeks (Q4W).
Period: Overall Study
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Started | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 5 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Site terminated by sponsor | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Death | 3 | 4 | 3 | 6 | 0 | 2 | 4 | 2 | 2 | 4 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W | Total
Number analyzed (Participants) | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.02) | 57.8 (15.41) | 62.3 (13.15) | 57.4 (12.57) | 67.0 (13.08) | 52.5 (10.08) | 67.0 (6.44) | 70.5 (12.02) | 68.0 (6.63) | 55.9 (10.61) | 62.9 (9.11) | 57.2 (13.86) | 70.0 (NA) — Could not be estimated due to insufficient number of participants | 60.8 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 5 | 1 | 3 | 4 | 1 | 3 | 4 | 4 | 1 | 0 | 33
  Male | 1 | 5 | 3 | 6 | 2 | 1 | 1 | 1 | 3 | 3 | 4 | 4 | 1 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Not Hispanic or Latino | 2 | 4 | 6 | 10 | 2 | 3 | 5 | 2 | 3 | 7 | 6 | 4 | 1 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 5
  White | 3 | 5 | 3 | 8 | 2 | 4 | 4 | 2 | 1 | 5 | 7 | 3 | 1 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A Dose-Limiting Toxicity (DLT) is defined as a treatment-related adverse event that meets specific severity criteria, excluding those clearly due to disease progression or unrelated causes. DLTs include: any Grade ≥3 non-hematologic toxicity (with exceptions like transient nausea, fatigue, rash, or electrolyte imbalances), significant liver enzyme elevations, Grade 4 neutropenia >7 days, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with bleeding, febrile neutropenia, and any Grade ≥3 immune-mediated toxicity including myocarditis, myelitis, or severe skin reactions. Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization.
Time Frame: From first dose (Day 1) till 28 days
Population: Participants were DLT evaluable if they received ≥75% of planned BMS-986408 doses without a DLT or had a DLT after at least one dose. In Part 2, they must also have received one nivolumab dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 4 | 6 | 9 | 3 | 3 | 4 | 2 | 2 | 3 | 8 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after signing of informed consent, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory test result), symptom, or disease temporally associated with the study intervention. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose (Day 1) till 30 days after the last dose (Up to approximately 13 months) for Group A to C and from Day 1 untill 100 days after last dose (up to approximately 15 months) for group D
Population: Safety population included all participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
Participants
  Any Adverse Events | 3 | 6 | 6 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
  Any Drug-related AEs | 2 | 4 | 3 | 11 | 3 | 4 | 4 | 2 | 3 | 6 | 6 | 5 | 1
  Serious Adverse Events | 2 | 1 | 2 | 7 | 2 | 3 | 4 | 2 | 4 | 3 | 3 | 3 | 1
  AEs leading to Discontinuation | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BMS-986408
Description: Blood samples were collected to assess pharmacokinetic parameters
Time Frame: Day 1 and 15 of Cycle 1 (Each cycle is of 28 days)
Population: PK evaluable population included all treated participants who have any available concentration-time data. Only participants with available concentration-time data at particular timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililitre (ng/mL)
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 5 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
nanogram per mililitre (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
  Cycle 1 Day 1 | 2.49 (61.05) | 4.86 (37.36) | 8.56 (35.16) | 15.00 (45.02) | 15.99 (64.67) | 5.57 (34.38) | 9.98 (21.58) | 11.20 (NA) — Not applicable as only 1 participant analyzed | 12.62 (37.65) | 19.43 (41.43) | 5.07 (36.26) | 10.71 (46.81) | 15.50 (NA) — Not applicable as only 1 participant analyzed
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 7 | 6 | 3 | 3 | 5 | 1 | 4 | 5 | 0 | 0 | 0
  Cycle 1 Day 15 | 9.32 (63.71) | 17.66 (36.70) | 22.19 (51.79) | 62.97 (80.05) | 41.27 (26.51) | 33.14 (61.85) | 67.55 (40.90) | 30.10 (NA) — Not applicable as only 1 participant analyzed | 28.43 (39.76) | 61.55 (32.92) |  |  |

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of BMS-986408
Description: Blood samples were collected to assess pharmacokinetic parameters
Time Frame: Day 1 and 15 of Cycle 1 (Each cycle is of 28 days)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 5 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
  Cycle 1 Day 1 | 2.52 (42.77) | 4.62 (23.00) | 4.22 (39.23) | 4.28 (43.77) | 5.38 (20.62) | 4.11 (3.08) | 3.57 (27.06) | 4.17 (NA) — Not applicable as only 1 participant analyzed | 3.19 (37.90) | 4.84 (21.23) | 3.90 (48.23) | 4.75 (22.10) | 5.97 (NA) — Not applicable as only 1 participant analyzed
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 7 | 6 | 3 | 3 | 5 | 1 | 4 | 5 | 0 | 0 | 0
  Cycle 1 Day 15 | 2.56 (90.49) | 4.02 (62.27) | 4.72 (89.13) | 3.12 (62.02) | 2.96 (115.92) | 3.71 (59.62) | 2.45 (28.62) | 2.10 (NA) — Not applicable as only 1 participant analyzed | 2.83 (41.44) | 4.14 (2.57) |  |  |

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration [AUC(0-T)]
Description: Blood samples were collected to assess pharmacokinetic parameters.
Time Frame: Day 1 and 15 of Cycle 1 (Each cycle is of 28 days)
Population: PK evaluable population included all treated participants who have any available concentration-time data. Only participants with with available concentration-time data at particular timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 5 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 7 | 11 | 3 | 3 | 5 | 1 | 6 | 7 | 8 | 5 | 1
  Cycle 1 Day 1 | 28.20 (195.49) | 78.06 (26.21) | 127.52 (37.45) | 190.26 (65.52) | 263.11 (46.78) | 21.59 (39.75) | 47.81 (25.65) | 45.09 (NA) — Not applicable as only 1 participant analyzed | 177.07 (37.21) | 275.58 (34.92) | 72.34 (26.97) | 132.88 (64.47) | 255.90 (NA) — Not applicable as only 1 participant analyzed
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 7 | 6 | 3 | 3 | 5 | 1 | 4 | 5 | 0 | 0 | 0
  Cycle 1 Day 15 | 188.79 (74.03) | 251.19 (83.24) | 435.29 (48.55) | 1252.68 (74.84) | 492.07 (124.61) | 178.12 (67.11) | 377.22 (38.40) | 170.18 (NA) — Not applicable as only 1 participant analyzed | 360.41 (132.44) | 736.15 (131.38) |  |  |

6. Secondary Outcome: Objective Response Rate (ORR) Per RECIST v1.1
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to the date of objectively documented progression per RECIST v1.1 or the date of subsequent anti-cancer therapy or death, whichever occurs first (up to approximately 12 months)
Population: Safety population included all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 84.2] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 97.5]

7. Secondary Outcome: Duration of Response Per RECIST v1.1
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death, whichever occurs first. Median computed using Kaplan-Meier method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 6
Population: Safety population included all participants who received at least 1 dose of study intervention. Only confirmed responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
months |  |  |  |  |  |  |  |  | NA [NA to NA] — Not estimable due to insufficient number of events. |  |  |  |

8. Primary Outcome: Number of Participants Who Died
Time Frame: From first dose (Day 1) until 100 days after the last dose (Up to approximately 15 months)
Population: Safety population included all participants who received at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
Number analyzed (Participants) | 3 | 6 | 7 | 11 | 3 | 4 | 5 | 2 | 6 | 7 | 8 | 5 | 1
Participants | 0 | 1 | 1 | 4 | 0 | 3 | 2 | 1 | 1 | 3 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from Day 1 and up to 107 weeks. Serious adverse events, other AEs were collected from first dose (Day 1) till 30 days after the last dose (Up to approximately 13 months) for Group A to C and from Day 1 until 100 days after last dose (up to approximately 15 months) for group D.
Description: Safety population included all participants who received at least 1 dose of study intervention.
Arm/Group | Part 1 (Group A) BMS-986408 0.75 mg QD | Part 1 (Group A) BMS-986408 1.5 mg QD | Part 1 (Group A) BMS-986408 3 mg QD | Part 1 (Group A) BMS-986408 5 mg QD | Part 1 (Group A) BMS-986408 7.25 mg QD | Part 1 (Group B) BMS-986408 1.5 mg BID | Part 1 (Group B) BMS-986408 2.25 mg BID | Part 1 (Group B) BMS-986408 3.75 mg BID | Part 1 Group C BMS-986408 3 mg QD | Part 1 Group C BMS-986408 5 mg QD | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/6 | 3/7 | 6/11 | 0/3 | 3/4 | 4/5 | 2/2 | 3/6 | 4/7 | 3/8 | 2/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/6 | 2/7 | 7/11 | 2/3 | 3/4 | 4/5 | 2/2 | 4/6 | 3/7 | 3/8 | 3/5 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/7 | 11/11 | 3/3 | 4/4 | 5/5 | 2/2 | 6/6 | 7/7 | 8/8 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Group A) BMS-986408 0.75 mg QD (N=3) | Part 1 (Group A) BMS-986408 1.5 mg QD (N=6) | Part 1 (Group A) BMS-986408 3 mg QD (N=7) | Part 1 (Group A) BMS-986408 5 mg QD (N=11) | Part 1 (Group A) BMS-986408 7.25 mg QD (N=3) | Part 1 (Group B) BMS-986408 1.5 mg BID (N=4) | Part 1 (Group B) BMS-986408 2.25 mg BID (N=5) | Part 1 (Group B) BMS-986408 3.75 mg BID (N=2) | Part 1 Group C BMS-986408 3 mg QD (N=6) | Part 1 Group C BMS-986408 5 mg QD (N=7) | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W (N=8) | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W (N=5) | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteric rupture (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Assisted suicide (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (Group A) BMS-986408 0.75 mg QD (N=3) | Part 1 (Group A) BMS-986408 1.5 mg QD (N=6) | Part 1 (Group A) BMS-986408 3 mg QD (N=7) | Part 1 (Group A) BMS-986408 5 mg QD (N=11) | Part 1 (Group A) BMS-986408 7.25 mg QD (N=3) | Part 1 (Group B) BMS-986408 1.5 mg BID (N=4) | Part 1 (Group B) BMS-986408 2.25 mg BID (N=5) | Part 1 (Group B) BMS-986408 3.75 mg BID (N=2) | Part 1 Group C BMS-986408 3 mg QD (N=6) | Part 1 Group C BMS-986408 5 mg QD (N=7) | Part 2 Group D BMS-986408 1.5 mg QD + NIVO 480 mg Q4W (N=8) | Part 2 Group D BMS-986408 3 mg QD + NIVO 480 mg Q4W (N=5) | Part 2 Group D BMS-986408 5 mg QD + NIVO 480 mg Q4W (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 3 | 2 | 1 | 2 | 0 | 1 | 4 | 0 | 3 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3 | 8 | 3 | 2 | 4 | 2 | 5 | 3 | 3 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 8 | 3 | 2 | 3 | 1 | 2 | 3 | 4 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 3 | 2 | 3 | 1 | 1 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 5 | 2 | 3 | 3 | 1 | 1 | 3 | 3 | 2 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 5 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinolaryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 2 | 1 | 4 | 4 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 3 | 3 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT05407675/Prot_SAP_000.pdf